CLINICAL TRIAL: NCT02440477
Title: The Effect of Changing Posture in Sitting on Selected Clinical Shoulder Tests in Patients With Rotator Cuff Degenerative Tears
Brief Title: The Effect of Changing Posture in Sitting on Selected Clinical Shoulder Tests
Acronym: EOCPIS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ק018/2015
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Partial Tear of Rotator Cuff

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- partial rotator cuff tears: 50 subjects with shoulder pain who are diagnosed with partial rotator cuff degenrative tears by ultrasound. All patients will be measured for their body weight and height and their hand dominance will be notified. Following reliability trials on the first 10 subjects, all subjects will be tested for pain provocation and level of pain (VAS) in both shoulders with 3 commonly used clinical shoulder tests for the diagnosis of rotator cuff diseases Empty can ,Neer test and Hawkins-Kennedy test in 3 sitting postures; normal resting posture, slouched posture, and upright posture with scapular retraction. In addition, the rotator cuff muscle strength tests during shoulder abduction, internal rotation and external rotation will be measured for the 2 shoulders using a hand-held dynamometer.
  Interventions: Other: clinical shoulder tests
- control group: 50 volunteering subjects without any pain in the upper quadrant.All patients will be measured for their body weight and height and their hand dominance will be notified. Following reliability trials on the first 10 subjects, all subjects will be tested for pain provocation and level of pain (VAS) in both shoulders with 3 commonly used clinical shoulder tests for the diagnosis of rotator cuff diseases Empty can ,Neer test and Hawkins-Kennedy test in 3 sitting postures; normal resting posture, slouched posture, and upright posture with scapular retraction. In addition, the rotator cuff muscle strength tests during shoulder abduction, internal rotation and external rotation will be measured for the 2 shoulders using a hand-held dynamometer.
  Interventions: Other: clinical shoulder tests

INTERVENTIONS:
Other: clinical shoulder tests — Three clinical shoulder tests (Neer impingement sign,Hawkins-kennedy, empty can) performed in three different sitting positions: normal resting posture, slouched posture, and upright posture with scapular retraction and shoulder. and in addition shoulder muscle strength test with handheld dynamometer

SUMMARY:
Background: Shoulder pain is the third most common musculoskeletal problem accounting almost 21% of all musculoskeletal complaints. Symptomatic Rotator cuff degenerative tears (RCDT) are mostly common above the age of 40. Deviations of posture in the upper quadrant such as, slouched posture and forward head position, have been linked repeatedly to rotator cuff diseases, altered scapular kinematics and changes in the acromiohumeral distance (AHD). No study yet examined the effect of changing posture in sitting on the output of shoulder clinical tests, in patients with RCDT.

Objectives: The primary objective of the study is to examine the effect of changing posture in sitting on selected clinical shoulder tests in patients with rotator cuff degenerative tears (RCDT) Study design: A single blinded controlled clinical trial Methods: A total of 100 subjects (Patients referred to physiotherapy outpatient clinics of Clalit Healthcare Services in Holon and Hertzlyia) will be included in this study and divided into 2 groups: 50 subjects with shoulder pain who are diagnosed with RCDT by ultrasound and a control group of 50 volunteering subjects without any pain in the upper quadrant. All patients will be measured for their body weight and height and their hand dominance will be notified. Following reliability trials on the first 10 subjects, all subjects will be tested for pain provocation and level of pain (VAS) in both shoulders with 3 commonly used clinical shoulder tests for the diagnosis of rotator cuff diseases (Empty can - sensitivity=94%, specificity = 46% Neer test - sensitivity = 72%, specificity = 60%, and Hawkins-Kennedy test - sensitivity = 79%, specificity = 59% ) in 3 sitting postures; normal resting posture, slouched posture, and upright posture with scapular retraction as described by Kalra et al (2010). In addition, the rotator cuff muscle strength tests during shoulder abduction, internal rotation and external rotation will be measured for the 2 shoulders using a hand-held dynamometer.

DETAILED DESCRIPTION:
Quality assurance - "clalit" health services will provide ongoing auditing and monitoring of the study. data checks will be also examined by "clalit health services". the investigators are obliged to enter all the data into logs provided upfront by the organisation. All the data obtained will be stored in an original folder intended for inspection and all encounters with volunteers will be documented in the computerized medical file of the volunteers. Standard operating procedures will be followed by the regulations expected by "clalit" health services and the Israeli ministry of health. After the first 10 volunteers of the study a reliability and validity statistical analysis will be made to assess the sample size estimated. Missing, unavailable, "non-reported" or uninterpretable data will be excluded from the final analysis.Data will be analyzed using the Statistical Package for the Social Sciences Version 15 (SPSS Inc., Chicago, IL, USA). Results of measurements of each test will be analyzed for mean, standard deviation (SD) and range. Categorical variables will be described percentiles/median. Changes of variables in the same subject will be analyzed using a paired T test for continuous variables and Mann-Whitney test for categorical variables. In addition, the correlations between variables will be calculated using ICC. P values smaller than 0.05 (p<0.05) will be considered significant

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 40 years.
2. Patients with partial rotator cuff degenerative tears that were diagnosed by ultrasound.

Exclusion Criteria:

1. Recent trauma to the upper quadrant.
2. Patients with spondyloarthropaties and or rheumatological diseases
3. Any oncological disease.
4. Any surgery or fractures in the upper quadrant.
5. Systemic vascular pathology.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged over 40 years with partial rotator cuff degenerative tears that were diagnosed by ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-07-01; Primary Completion 2017-04-01 (Estimated); Study Completion 2017-04-01 (Estimated)

PRIMARY OUTCOMES:
Neer test , empty can test, Hawkins Kennedy test | one year

SECONDARY OUTCOMES:
shoulder muscle testing | one year

CONTACTS AND LOCATIONS:
Overall Officials: shlomo bierkenfeld, MD, Principal Investigator — Clalit Health Services
Locations (2):
- Israel (2):
  - Bat yamon physical therapy, Bat Yam, Israel
  - Holon Physiotherapy, Holon, Israel

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Urwin M, Symmons D, Allison T, Brammah T, Busby H, Roxby M, Simmons A, Williams G. Estimating the burden of musculoskeletal disorders in the community: the comparative prevalence of symptoms at different anatomical sites, and the relation to social deprivation. Ann Rheum Dis. 1998 Nov;57(11):649-55. doi: 10.1136/ard.57.11.649. PMID 9924205
- [Background] Kalra N, Seitz AL, Boardman ND 3rd, Michener LA. Effect of posture on acromiohumeral distance with arm elevation in subjects with and without rotator cuff disease using ultrasonography. J Orthop Sports Phys Ther. 2010 Oct;40(10):633-40. doi: 10.2519/jospt.2010.3155. PMID 20710092
- [Background] Bullock MP, Foster NE, Wright CC. Shoulder impingement: the effect of sitting posture on shoulder pain and range of motion. Man Ther. 2005 Feb;10(1):28-37. doi: 10.1016/j.math.2004.07.002. PMID 15681266
- [Background] Cutti AG, Veeger HE. Shoulder biomechanics: today's consensus and tomorrow's perspectives. Med Biol Eng Comput. 2009 May;47(5):463-6. doi: 10.1007/s11517-009-0487-3. Epub 2009 Apr 25. PMID 19396486
- [Background] Lugo R, Kung P, Ma CB. Shoulder biomechanics. Eur J Radiol. 2008 Oct;68(1):16-24. doi: 10.1016/j.ejrad.2008.02.051. Epub 2008 Jun 3. PMID 18511227
- [Background] Lewis JS. Subacromial impingement syndrome: a musculoskeletal condition or a clinical illusion? Physical Therapy Reviews.2011; 16(5): 1-12.
- [Background] Kebaetse M, McClure P, Pratt NA. Thoracic position effect on shoulder range of motion, strength, and three-dimensional scapular kinematics. Arch Phys Med Rehabil. 1999 Aug;80(8):945-50. doi: 10.1016/s0003-9993(99)90088-6. PMID 10453773
- [Background] Donatelli R. Physical Therapy of the Shoulder (Clinics in Physical Therapy). 4th ed. New York, NY: Churchill-Livingstone; 2004.
- [Background] Neer CS 2nd. Impingement lesions. Clin Orthop Relat Res. 1983 Mar;(173):70-7. No abstract available. PMID 6825348
- [Background] Greenfield B, Catlin PA, Coats PW, Green E, McDonald JJ, North C. Posture in patients with shoulder overuse injuries and healthy individuals. J Orthop Sports Phys Ther. 1995 May;21(5):287-95. doi: 10.2519/jospt.1995.21.5.287. PMID 7787853
- [Background] Culham E, Peat M. Functional anatomy of the shoulder complex. J Orthop Sports Phys Ther. 1993 Jul;18(1):342-50. doi: 10.2519/jospt.1993.18.1.342. PMID 8348135
- [Background] Ludewig PM, Reynolds JF. The association of scapular kinematics and glenohumeral joint pathologies. J Orthop Sports Phys Ther. 2009 Feb;39(2):90-104. doi: 10.2519/jospt.2009.2808. PMID 19194022
- [Background] Lukasiewicz AC, McClure P, Michener L, Pratt N, Sennett B. Comparison of 3-dimensional scapular position and orientation between subjects with and without shoulder impingement. J Orthop Sports Phys Ther. 1999 Oct;29(10):574-83; discussion 584-6. doi: 10.2519/jospt.1999.29.10.574. PMID 10560066
- [Background] Hegedus EJ, Goode A, Campbell S, Morin A, Tamaddoni M, Moorman CT 3rd, Cook C. Physical examination tests of the shoulder: a systematic review with meta-analysis of individual tests. Br J Sports Med. 2008 Feb;42(2):80-92; discussion 92. doi: 10.1136/bjsm.2007.038406. Epub 2007 Aug 24. PMID 17720798
- [Background] Schellingerhout JM, Verhagen AP, Thomas S, Koes BW. Lack of uniformity in diagnostic labeling of shoulder pain: time for a different approach. Man Ther. 2008 Dec;13(6):478-83. doi: 10.1016/j.math.2008.04.005. Epub 2008 Jun 13. PMID 18555732
- [Background] Hughes PC, Taylor NF, Green RA. Most clinical tests cannot accurately diagnose rotator cuff pathology: a systematic review. Aust J Physiother. 2008;54(3):159-70. doi: 10.1016/s0004-9514(08)70022-9. PMID 18721119
- [Background] Tempelhof S, Rupp S, Seil R. Age-related prevalence of rotator cuff tears in asymptomatic shoulders. J Shoulder Elbow Surg. 1999 Jul-Aug;8(4):296-9. doi: 10.1016/s1058-2746(99)90148-9. PMID 10471998
- [Background] Lewis JS, Tennent TD. How effective are diagnostic tests for the assessment of rotator cuff disease of the shoulder? In: MacAuley D, Best TM, editors. Evidence based Sports Medicine. 2nd ed. London: Blackwell Publishing. 2007; 327-59.
- [Background] Jobe FW, Moynes DR. Delineation of diagnostic criteria and a rehabilitation program for rotator cuff injuries. Am J Sports Med. 1982 Nov-Dec;10(6):336-9. doi: 10.1177/036354658201000602. PMID 7180952
- [Background] Hawkins RJ, Kennedy JC. Impingement syndrome in athletes. Am J Sports Med. 1980 May-Jun;8(3):151-8. doi: 10.1177/036354658000800302. PMID 7377445
- [Background] Kim E, Jeong HJ, Lee KW, Song JS. Interpreting positive signs of the supraspinatus test in screening for torn rotator cuff. Acta Med Okayama. 2006 Aug;60(4):223-8. doi: 10.18926/AMO/30715. PMID 16943859
- [Background] Michener LA, Kalra N, Pinkstaff S, Ericksen J,Boardman N. Measurement of the subacromial space using ultrasonography. Journal of Athletic Training.2007;42:126.
- [Background] Woo S.L. An K.N. Frank C.B. Livesay G.A. Ma, C.B. Zeminski J. Anatomy, biology, and biomechanics of tendon and ligament. 2000 In: Buckwalter, J., Einhorn, T.,Simon, S. (Eds.), Orthopaedic Basic Science. American Academy of Orthopaedic Surgeons, Park Ridge.
- [Background] Kumagai J, Sarkar K, Uhthoff HK. The collagen types in the attachment zone of rotator cuff tendons in the elderly: an immunohistochemical study. J Rheumatol. 1994 Nov;21(11):2096-100. PMID 7869316
- [Background] Seitz AL, McClure PW, Finucane S, Boardman ND 3rd, Michener LA. Mechanisms of rotator cuff tendinopathy: intrinsic, extrinsic, or both? Clin Biomech (Bristol). 2011 Jan;26(1):1-12. doi: 10.1016/j.clinbiomech.2010.08.001. Epub 2010 Sep 16. PMID 20846766
- [Background] Palstanga N, Field D, Soamnes R. Anatomy and human movement, structure and function, third edition. Butterworth-Heinman Ltd. 1991: 88-101
- [Background] Magee DJ. Orthopedic Physical Assessment: 5th Edition. St. Louis, MO: Saunders Elsevier; 2008.
- [Background] Kendall FP, Kendall McCreary E, Rodgers MM, Romani WA. Muscles: Testing and Function, with Posture and Pain 5th edition. LWW; 2005.
- [Derived] Weisman A, Masharawi Y. Does Altering Sitting Posture Have a Direct Effect on Clinical Shoulder Tests in Individuals With Shoulder Pain and Rotator Cuff Degenerative Tears? Phys Ther. 2019 Feb 1;99(2):194-202. doi: 10.1093/ptj/pzy111. PMID 30351428